CLINICAL TRIAL: NCT00673686
Title: Single Center, Double-blind, Randomized Study to Compare the Effect of SH T 00186 D on Follicular Development in a 24-day Regimen Versus a 21-day Regimen in Healthy Female Volunteers
Brief Title: Study to Investigate the Effect of Missed Pills on Follicular Development in Two Application Regimens of SH T 00186 D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91377; 308382
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Contraceptives, Oral
Keywords: Oral contraceptive; Ovulation; Missing pills; Intake compliance; Cycle control
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; drospirenone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Active Comparator)
  Interventions: Drug: Yasminelle (SH T 00186 D)
- Arm 1 (Experimental)
  Interventions: Drug: YAZ (DRSP 3 mg/EE 0.02 mg, BAY86-5300)

INTERVENTIONS:
Drug: YAZ (DRSP 3 mg/EE 0.02 mg, BAY86-5300) — SH T 00186 D in a 24-day regimen, i.e., 24 verum tablets, 4 placebo tablets Dose: 0.02 mg EE, 3 mg DRSPMode of administration: Oral, 1 tablet dailyDuration of treatment: 3 cycles of 28 days each
  Arms: Arm 1
Drug: Yasminelle (SH T 00186 D) — SH T 00186 D in a 21-day regimen, i.e., 21 verum tablets, 7 placebo tablets Dose: 0.02 mg EE, 3 mg DRSPMode of administration: Oral, 1 tablet dailyDuration of treatment: 3 cycles of 28 days each
  Arms: Arm 2

SUMMARY:
In this study a comparison was made on the influence of missing pills on follicular ripening. By missing a given number of pills, an effect on "contraceptive robustness" of the two investigated contraceptive pills was measured by ultrasound comparison of follicular size and other parameters which indicate how far ovulation might be.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18 to 35 years inclusive (smokers aged up to 30 years inclusive)
* No contraindications for combined oral contraceptive (COC) use
* Follicular diameter of greater-equal than 15 mm on visit 6 (admission to treatment), or an observed ovulation during pretreatment cycle Exclusion Criteria:
* Pregnancy or lactation- Substantial overweight, i.e., body mass index (BMI) > 30,
* Known hypersensitivity to any of the study drug ingredients
* Any disease that may worsen under hormonal treatment or might interfere with the conduct of the study, or the interpretation of the results

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2004-05; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Hoogland scores in cycles 2 and 3 | Treatment cycles 2 and 3 (treatment weeks 5-12)

SECONDARY OUTCOMES:
Follicle size | Treatment cycles 2 and 3 (treatment weeks 5-12
Hormone levels of progesterone, estradiol, luteinizing hormone, follicle stimulating hormone | Treatment cycles 2 and 3 (treatment weeks 5-12
Endometrial thickness | Treatment cycles 2 and 3 (treatment weeks 5-12
Cervical mucus | Treatment cycles 2 and 3 (treatment weeks 5-12

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Groningen, Netherlands

REFERENCES:
- [Result] Anttila L, Neunteufel W, Petraglia F, Marr J, Kunz M. Cycle control and bleeding pattern of a 24/4 regimen of drospirenone 3 mg/ethinylestradiol 20 mug compared with a 21/7 regimen of desogestrel 150 mug/ethinylestradiol 20 mug: a pooled analysis. Clin Drug Investig. 2011;31(8):519-525. doi: 10.2165/11590260-000000000-00000. PMID 21721590